CLINICAL TRIAL: NCT04852965
Title: Early Detection of Late Anthracycline Induced Cardiotoxicity in Survivors of Childhood Malignancy
Brief Title: Late Anthracycline Induced Cardiotoxicity- Childhood Cancer Survivors
Status: Active, not recruiting | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Chris Watson, Senior Lecturer, Queen's University, Belfast
Other Study IDs: B21/01
Record Dates: First submitted 2021-04-01; First posted 2021-04-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anthracycline Induced Cardiotoxicity
Keywords: Anthracycline; Doxorubicin; Cardiotoxicity; Strain; IL6; sST2; MPO; Cardiomyopathy; Transcriptomics; MRI; Echocardiography; Cardio-oncology; Proteomics
MeSH Terms: conditions — Cardiotoxicity; Sprains and Strains; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be collected for currently used (for example troponin, NTproBNP,) and novel (for example, IL6, MPO, and sST2) biomarkers to see if we can predict early cardiomyopathy. Transcriptomics and proteomics based biomarker discovery will identify new biomarkers to allow timely diagnosis.
Oversight: Data Monitoring Committee: No

SUMMARY:
Anthracyclines treat up to 60% of childhood malignancies with remarkable improvements survival rates. Unfortunately anthracyclines are associated with an increased cardiomyopathy risk. One study showed an almost six-fold greater risk of developing cardiomyopathy compared to sibling controls. A retrospective pilot study showed evidence of subclinical dysfunction (including impaired global longitudinal strain) in 42/52 childhood cancer survivors. There is limited research in this area, therefore current guidelines are based on expert opinion alone and lack consensus. Current methods of detection diagnose cardiomyopathy at an irreversible stage i.e. when the compensatory mechanisms are exhausted and the left ventricular ejection fraction impaired. Small trials have shown that early treatment with standard heart failure therapy may reverse damage, further validation is however required in this cohort.

Newer techniques such as tissue doppler and strain rate imaging have shown promise for early prediction of cardiomyopathy in adult studies. Biomarkers such as troponin and NT-proBNP have also shown a correlation with cardiomyopathy.

This study (n=208) aims to use echocardiography, strain imaging, holter monitoring and MRI for early detection of cardiomyopathy. Biomarkers, both currently used (for example, troponin and NTproBNP,) and more novel (for example, IL6, MPO, and sST2) will be assessed to see if early cardiomyopathy can be predicted.

This study will explore biomarker discovery by analysing an age/gender matched subgroup for the top differentially expressed microRNA and protein biomarkers. Selected biomarkers will then be validated in a larger cohort.

DETAILED DESCRIPTION:
CLINICAL APPOINTMENT A linked anonymised Case Report Form will be completed using participant answers and relevant aspects of their electronic care record. This will involve questions about the patient's demographics, chemotherapy history, cardiac symptoms, past medical history, medication history and family history.

Consenting patients will then have

* height, weight and blood pressure taken
* cardiovascular and respiratory examination Participants will then undergo
* SF36 quality of life questionnaire
* 6 minute walk test, grip strength
* Electrocardiogram by a trained researcher
* Venesection- 40ml blood sample from a peripheral vein by the trained researcher Crevicular fluid sample

INVESTIGATIONS

Participants will be invited for:

1. 24 hour holter monitor- arrhythmia assessment
2. Echocardiogram- diastolic and systolic function assessment, valvular analysis, global longitudinal strain
3. Magnetic resonance imaging (MRI) scan of the heart- volumetric analysis, late gadolinium enhancement and STIR imaging assessments. As part of the scan the patient will require a venflon to be inserted into a peripheral vein for gadolinium injection. A safety questionnaire will be sent to the patient prior to attendance as part of standard MRI procedure. All safety aspects will be re-assessed on the day of attendance by a trained radiographer

BLOOD SAMPLE ANALYSIS Blood samples will be sent for standard of care and cardiovascular risk assessment. Tests include a full blood picture, urea and electrolytes, C-reactive protein, iron profile, B12 and folate, lipid profile, HbA1c, NT-proBNP and high sensitivity troponin.

Additional disease associated biomarkers for example sST2, MPO, and IL6 will be quantified using immunoassays. Biomarker discovery, including transcriptomics and proteomics will be carried out to identify signatures that could predict cardiotoxicity, subclinical dysfunction, and cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

-Male and female patients over the age of 18 who have received at least moderate (100mg/m2) anthracycline chemotherapy as a child (<16 years).

Exclusion Criteria:

* patients born with complex heart disease
* patients who would not be safely able to have a magnetic resonance imaging scan
* patients who cannot give consent
* patients under the age of 18 or who have had less than a moderate dose of anthracycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients identified by paediatric oncology who have received anthracycline therapy in childhood.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity | 2 years
  Number of participants with anthracycline related cardiotoxicity as defined by the British Society of Echocardiography and British Cardio-Oncology Society guidelines

SECONDARY OUTCOMES:
Incidence of myocardial injury | 2 years
  Levels of high sensitivity troponin T and NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: Lana J Dixon, MB BCh BAO, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Belfast Health and Social Care Trust, Belfast, United Kingdom

REFERENCES:
- [Background] Thompson KA. Pregnancy and Cardiomyopathy After Anthracyclines in Childhood. Front Cardiovasc Med. 2018 Mar 26;5:14. doi: 10.3389/fcvm.2018.00014. eCollection 2018. PMID 29632865
- [Background] Mulrooney DA, Yeazel MW, Kawashima T, Mertens AC, Mitby P, Stovall M, Donaldson SS, Green DM, Sklar CA, Robison LL, Leisenring WM. Cardiac outcomes in a cohort of adult survivors of childhood and adolescent cancer: retrospective analysis of the Childhood Cancer Survivor Study cohort. BMJ. 2009 Dec 8;339:b4606. doi: 10.1136/bmj.b4606. PMID 19996459
- [Background] Curigliano G, Cardinale D, Suter T, Plataniotis G, de Azambuja E, Sandri MT, Criscitiello C, Goldhirsch A, Cipolla C, Roila F; ESMO Guidelines Working Group. Cardiovascular toxicity induced by chemotherapy, targeted agents and radiotherapy: ESMO Clinical Practice Guidelines. Ann Oncol. 2012 Oct;23 Suppl 7:vii155-66. doi: 10.1093/annonc/mds293. PMID 22997448
- [Background] Cardinale D, Colombo A, Lamantia G, Colombo N, Civelli M, De Giacomi G, Rubino M, Veglia F, Fiorentini C, Cipolla CM. Anthracycline-induced cardiomyopathy: clinical relevance and response to pharmacologic therapy. J Am Coll Cardiol. 2010 Jan 19;55(3):213-20. doi: 10.1016/j.jacc.2009.03.095. PMID 20117401
- [Background] Sawaya H, Sebag IA, Plana JC, Januzzi JL, Ky B, Tan TC, Cohen V, Banchs J, Carver JR, Wiegers SE, Martin RP, Picard MH, Gerszten RE, Halpern EF, Passeri J, Kuter I, Scherrer-Crosbie M. Assessment of echocardiography and biomarkers for the extended prediction of cardiotoxicity in patients treated with anthracyclines, taxanes, and trastuzumab. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):596-603. doi: 10.1161/CIRCIMAGING.112.973321. Epub 2012 Jun 28. PMID 22744937
- [Background] Cardinale D, Sandri MT, Colombo A, Colombo N, Boeri M, Lamantia G, Civelli M, Peccatori F, Martinelli G, Fiorentini C, Cipolla CM. Prognostic value of troponin I in cardiac risk stratification of cancer patients undergoing high-dose chemotherapy. Circulation. 2004 Jun 8;109(22):2749-54. doi: 10.1161/01.CIR.0000130926.51766.CC. Epub 2004 May 17. PMID 15148277
- [Background] Romano S, Fratini S, Ricevuto E, Procaccini V, Stifano G, Mancini M, Di Mauro M, Ficorella C, Penco M. Serial measurements of NT-proBNP are predictive of not-high-dose anthracycline cardiotoxicity in breast cancer patients. Br J Cancer. 2011 Nov 22;105(11):1663-8. doi: 10.1038/bjc.2011.439. Epub 2011 Nov 8. PMID 22068815